CLINICAL TRIAL: NCT06833580
Title: Effects of a Health Belief Model-Based Fall Prevention Education Program on Health Literacy and Physical Function in Patients With Chronic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Nuha Awadh Alharbi, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E-24-9164
Record Dates: First submitted 2025-02-17; First posted 2025-02-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-02

CONDITIONS: Fall Prevention; Chronic Stroke Patients; Health Literacy; Education of Patients; Health Belief Model

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (receive the health belief model-based fall prevention education program) (Experimental): Each participant in this group will receive two in-person individual educational sessions based on the health belief model (HBM)
  Interventions: Other: The intervention group, who will receive the health belief model-based fall prevention education program
- The control group, who will receive their usual intervention in the physical therapy clinic (No Intervention): Each participant in this group will receive their usual intervention in the physical therapy clinic

INTERVENTIONS:
Other: The intervention group, who will receive the health belief model-based fall prevention education program — Each participant in this group will receive two in-person individual educational sessions based on the health belief model (HBM).
  Arms: The intervention group (receive the health belief model-based fall prevention education program)

SUMMARY:
The goal of this clinical trial is to to evaluate the effects of a health belief model-based fall prevention education program on health literacy and physical function, fall rate, fall risk, fear of fall, and quality of life in patients with chronic stroke.

The main question it aim to answer is

* Does a health belief model-based fall prevention education program have a positive effect on health literacy, physical function, fall risk, fear of falling, and quality of life in patients with chronic stroke?

Researchers will compare the intervention group, who will receive the health belief model-based fall prevention education program, to the control group, who will receive their usual intervention in the physical therapy clinic, to see if the health belief model-based fall prevention education program has an effect on health literacy and physical function, fall rate, fall risk, fear of falling, and quality of life in patients with chronic stroke.

The clinical trial will be conducted in four phases; each participant will take around 6 weeks and will receive two in-person individual educational sessions based on the health belief model (HBM).

ELIGIBILITY:
Inclusion Criteria:

* Aged 45 years and older
* Diagnosed with stroke (more than 6 months),
* No cognitive impairment (Arabic version of Mini-Mental State Examination [MMSE-A] score of 24 or more)
* No visual or hearing impairment
* Able to walk independently or with assistive devices for 10 meters

Exclusion Criteria:

* Severe communication deficiencies.
* Having neurological conditions other than stroke or other serious medical conditions that precluded participation in the study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-03-12 (Estimated)

PRIMARY OUTCOMES:
European Health Literacy Survey (HLS-EU-Q16) | Before and after intervention and one month after the intervention
  The Arabic version of the European Health Literacy Survey Questionnaire (Ar- HLS-EU) will be used to assess health literacy (HL).
  It is a self-reported questionnaire that consists of 16 items that measure the individual's ability to access, understand, process, and apply health information.
  Each respondent expresses an opinion on a specific statement on the Likert 4-point scale (very easy, easy, difficult, very difficult).
  The responses are dichotomized into easy (given a value of 1) and difficult (given a value of 0).
  Total scores range from 0 to 16, in which zero represented the lowest possible HL and 16 represented the highest possible one. Then, participants' scores were categorized into inadequate (0-8), problematic (9-12), and sufficient (13-16) health literacy.
  The HLS-EU-Q16 has been translated to the Arabic language and reported to be valid and reliable.
Falls Risk Questionnaire (FRQ) | Before and after intervention and one month after the intervention
  FRQ is a self-reported questionnaire used to assess personal fall risk awareness. It contains 12 yes/no questions assessing different fall- risk factors in older adults.
  The answers were scored as (No = 0) or (Yes = 2) for the first two questions and (Yes = 1) for the remaining 10 questions.
  Individuals scoring four or more were considered at increased risk of falling. The Arabic version of FRQ It is highly valid and reliable in providing valuable data for evaluating fall risk.
The Iconographical Falls Efficacy Scale - Short Version (Icon-FES) | Before and after intervention and one month after the intervention
  Short Version of Icon-FES will be used to assess concern about falling during 10 activities of daily living through a combination of images and brief descriptions.
  Participants will be instructed to carefully observe each image and visualize themselves performing the activity.
  Each item is rated on a 4-point scale (1 = not at all concerned to 4 = very concerned), with facial expression icons providing a visual representation of concern levels.
  The total Icon-FES score ranges from 10 to 40, where 10-18 indicates low concern about falling, and 19-40 reflects high concern.
  The Arabic short version of Icon-FES has been proven to be a reliable and valid tool for assessing fall-related concern in community-dwelling older adults.

SECONDARY OUTCOMES:
Five Times Sit-To-Stand (5TSTS) | Before and after intervention and one month after the intervention
  5TSTS will be used to assess functional lower extremity strength. It measured the time (in seconds) taken to complete 5 repetitions of the sit-to-stand from a seated position.
  To perform the test, the patient sits in a standardized chair (height 43 cm and depth 47.5 cm), with arms crossed over his chest and with his back resting on the back of the chair.
  The patients were instructed to stand up and sit down five times as fast as possible with the command "GO." The patient had to stand fully between repetitions of the test and not touch the back of the chair during each repetition. Timing began at "GO" and ended when the patient's back touched the backrest of the chair after the fifth repetition The shorter the time taken by the patient, the better their functional condition. 5STS is valid and has an excellent intraclass correlation coefficient (ICC) (range,.970-.976) in patients with chronic stroke
Time Up and Go (TUG) | Before and after intervention and one month after the intervention
  TUG will be used to measure functional mobility and balance in a short time. The test involved standing up from a chair, walking 3 meters, turning, walking back to the chair, and sitting down.
  Participants were allowed to use their walking aid and to use the armrest for support when getting up. The time will be recorded in seconds from standing up to sitting down.
  TUG will be performed twice and the mean of the 2 trials will be used. A shorter time indicates better functional mobility. Patients who take ≥14 seconds to complete the TUG are at risk for falling.
  TUG has been reported to have excellent test-retest reliability (ICC = 0.95-0.97) in patients with chronic stroke.
Stroke Specific Quality of Life Scale - Short Version (SS-QOL) | Before and after intervention and one month after the intervention
  A short version of the Stroke Specific Quality of Life Scale will be used to assess quality of life. The SS-QOL-12-AR adopts a two-domain structure and incorporates 12 selected items derived from the original 49-item SSQOL-A scale.
  The psychosocial domain includes seven items involving thinking, family roles, social roles, personality, mood, energy, and language. Additionally, the physical domain comprises five items addressing self-care, mobility, upper extremity function, vision, and work.
  Each of the 12 items is assessed using a consistent five-point scale that aligns with its corresponding item in the original SSQOL-A scale.
  Responses from each item are summed up, and the resulting composite score ranges from a minimum of 12 to a maximum of 60, with higher scores indicating a better QOL. The SS-QOL-12 has been translated to Arabic and it has excellent psychometric properties.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Sultan military medical city, Riyadh, Riyadh Region, Saudi Arabia